CLINICAL TRIAL: NCT02343393
Title: Nitrates In Combination With Hydralazine in cardiorEnal Syndrome (NICHE) Study
Acronym: NICHE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Singapore Clinical Research Institute (Other); Changi General Hospital (Other); National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NICHE
Record Dates: First submitted 2015-01-15; First posted 2015-01-22 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Cardio-Renal Syndrome
Keywords: Endothelial Dysfunction; Biomarkers; Hydralazine-Isosorbide Dinitrate
MeSH Terms: conditions — Cardio-Renal Syndrome | interventions — Hydralazine; Isosorbide Dinitrate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- H-ISDN (Experimental): Eligible patients randomised to treatment arm will be initiated on a starting dose of hydralazine 60mg and ISDN 30mg daily (20/10mg three times daily). After 7 days following the first dose, if the starting medication is well-tolerated, the patient is instructed to double the dose of study medication to the target maintenance dose of hydralazine 120mg and ISDN 60mg daily for 24 weeks
  Interventions: Drug: Hydralazine; Drug: Isosorbide Dinitrate
- Standard Medical Therapy (No Intervention): Current standard HF therapy include the use of beta-blockers, ACE inhibitors/ARBs and diuretics.

INTERVENTIONS:
Drug: Hydralazine
  Arms: H-ISDN
Drug: Isosorbide Dinitrate
  Arms: H-ISDN

SUMMARY:
This is a single-blind, randomised, clinical trial assessing the efficacy of Hydralazine and Isosorbidedinitrate combination (oral agents) in HF patients with renal dysfunction.

DETAILED DESCRIPTION:
Cardiorenal syndrome (CRS), where renal failure and heart failure (HF) co-exist in a vicious cycle, is a very common problem of great morbidity and mortality. The management of CRS is challenging as therapeutic options are mutually contradictory and largely empirical.

Endothelial dysfunction from oxidative injury has recently emerged as a common link between the failing heart and kidneys in CRS. The endothelium plays an obligatory role in cardiovascular homeostasis, and impaired endothelium-mediated nitric oxide (NO) bioavailability is the hallmark of endothelial dysfunction. There is a high prevalence of endothelial dysfunction in our Asian HF patients, with a greater degree of dysfunction seen in those with CRS. We hypothesise that targeting endothelial dysfunction may improve clinical status among Asian patients with CRS.

Isosorbide dinitrate (ISDN) increases NO bioavailability. Concomitant hydralazine (H) therapy prevents nitrate tolerance and protects NO from oxidative stress-induced degradation. The synergistic combination of H-ISDN is thought to exert beneficial effects on the endothelium.

We aim to perform a prospective randomised controlled trial to assess the effect of H-ISDN therapy for 6 months on exercise capacity, endothelial function, renal function, clinical outcomes and quality of life (QOL) in Asian patients with CRS. Specifically, we hypothesise that H-ISDN therapy will lead to improvement in exercise capacity (6 minute walk test (6MWT)), endothelial dysfunction (assessed by non-invasive peripheral arterial tonometry(PAT)), renal function, cardiac structure and function, clinical outcomes (all-cause mortality, HF hospitalisations) and QOL in Asian patients with CRS.

ELIGIBILITY:
Inclusion Criteria:

1. At least 21 years of age
2. Asian patients with symptomatic HF (regardless of EF) and renal impairment (eGFR<60ml/min/1.73m2)
3. At least one hospitalisation for HF during the preceeding year
4. On stable (at least 1 month) optimal medical therapy (maximum tolerated doses of ACE inhibitors or ARBs, beta blockers and aldosterone antagonists for HFREF, and optimally managed cardiovascular risk factors for HFPEF)
5. Able to complete 6 minute walk test (6MWT)
6. Able to maintain a systolic blood pressure ≥100mmHg
7. Able to provide written informed consent

Exclusion Criteria:

1. On chronic therapy with hydralazine and/or nitrates.
2. Known hypersensitivity to hydralazine and/or nitrates
3. Concurrent use of phosphodiesterase type 5 (PDE5) inhibitors
4. Females who are pregnant, nursing, or of childbearing potential and not practising effective contraception
5. Have had acute myocardial infarction, unstable or stable angina pectoris, or a cerebrovascular accident within the last 3 months
6. Have had cardiac revascularisation within the last 3 months or are likely to require coronary revascularisation within the study period
7. Have had cardiac arrest or life-threatening ventricular arrhythmia requiring intervention within 3 months
8. Rapidly deteriorating HF (2 admissions for acute decompensated HF, not due to non-compliance, within 6 months)
9. eGFR< 15ml/min/1.73m2, or on regular dialysis, or planned dialysis within the study period
10. Serious medical condition, emergency condition, uncontrolled systemic disease or any other medical condition that, in the judgement of the investigator, prohibits the patient from entering or potentially completing the study
11. Planned participation in any other interventional study or having received trial medication in the last 4 weeks within a clinical trial

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Effort tolerance by assessing 6 Minute Walk Test (6MWT) | 24 weeks

SECONDARY OUTCOMES:
Endothelial function as measured via a reactive hyperaemic index (RHI) by Peripheral Arterial Tonometry (PAT) | 24 weeks
Renal function (eGFR, Cystatin C, markers of kidney injury (proteinuria as quantified by urine protein-creatinine ratio (uPCR), NGAL)) | 24 weeks
Cardiac structure and function by 2D and Doppler echocardiography | 24 weeks
Quality of Life by self-reported 36-item Short Form Health Survey (SF-36) | 24 weeks
Clinical outcomes by recording deaths and HF hospitalisations | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Su Ping Carolyn Lam, MBBS, MRCP, MS, Study Chair — National University Hospital, Singapore
Locations (3):
- Singapore (3):
  - National University Hospital, Singapore, Singapore
  - National Heart Centre Singapore, Singapore
  - Changi General Hospital, Singapore